CLINICAL TRIAL: NCT04661306
Title: Optimizing Efficiency and Impact of Internet-delivered Insomnia Treatment for Cancer Caregivers
Brief Title: The Better Sleep for Supporters With Insomnia Study
Acronym: BeSSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kelly Shaffer, PhD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3809
Record Dates: First submitted 2020-10-28; First posted 2020-12-10 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Family Caregivers; Cancer; Insomnia; Sleep Initiation and Maintenance Disorders
Keywords: Family Caregivers; Cancer; Insomnia
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHUTi (Experimental)
  Interventions: Behavioral: SHUTi (Sleep Healthy Using the Internet)

INTERVENTIONS:
Behavioral: SHUTi (Sleep Healthy Using the Internet) — Cognitive Behavioral Therapy for insomnia delivered online and metered out over 6 weeks in a fully automated, interactive, tailored web-based program
  Other Names: CBTi

SUMMARY:
This study will identify whether - and if so, how - tailoring would increase adoption of and benefit from an interactive internet intervention for insomnia called SHUTi (Sleep Healthy Using the Internet) for cancer caregivers. Participating caregivers' sleep and sleep-related characteristics will be characterized from a baseline assessment; then, caregivers will receive complementary and voluntary access to SHUTi. Among caregivers who choose to use SHUTi, intervention use, perceived appropriateness, and effects on sleep and quality of life will be assessed. Among caregivers who choose not to use SHUTi, reasons and barriers to using the intervention will be assessed.

DETAILED DESCRIPTION:
Insomnia is a significant public health problem with substantial medical, psychological and financial ramifications. About 50-75% of the 3.5 million Americans who provide unpaid medical, practical, and/or emotional support for a loved one with cancer endorse clinically significant sleep disturbance. Understanding caregivers' psychosocial risk factors and needs, and the extent to which these are unique to the cancer caregiving context, will ensure appropriate and effective interventions for cancer caregivers with insomnia.

Existing psychosocial services for caregivers are primarily delivered in-person. Although such interventions are effective, they suffer from low enrollment, high dropout, and limited reach to caregivers who already have inadequate healthcare access, like caregivers from lower SES or those in rural areas. Digital health interventions can lower barriers to entry to supportive care for caregivers as they are conveniently accessible anywhere and anytime from an Internet-enabled device. Sleep Healthy Using the Internet (SHUTi) is a NCI-designated research-tested intervention that delivers cognitive-behavioral therapy for insomnia (CBT-I) and holds significant potential to accessibly treat insomnia for cancer caregivers. Most digital health interventions tested among caregivers, however, have been developed de novo for specific caregiving contexts. The implicit assumption underlying highly tailored interventions for caregivers is that caregivers have different deficits, risk factors, and needs from non-caregivers. This assumption has not often been tested, and therefore the extent to which caregivers want and need tailoring for digital health interventions is not known. This study is therefore designed to provide the data necessary to ensure the highest quality, impact, and efficiency from existing evidence-based digital health interventions to meet pressing psychosocial needs among cancer caregivers. Specifically, this study will directly inform next research steps for tailoring and testing SHUTi for optimal impact and reach among caregivers.

The SHUTi Program: SHUTi is a self-guided (i.e., automated), interactive, and tailored web-based program modeled on the primary tenants of face-to-face CBT-I (sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, relapse prevention). Intervention content is metered out over time through 6 "Cores." Users obtain access to a new Core based on a time and event-based schedule (e.g., 7 days after completion of previous Core). This schedule is consistent with the recommendation from a task force commissioned by the Academy of Sleep Medicine, which deemed that an average of 6 - 8 sessions constitutes "adequate treatment exposure". The SHUTi program relies on user-entered online Sleep Diaries to track progress and to tailor treatment recommendations (i.e., assign a "sleep restriction" window). Each Core acts as an online analog for the weekly sessions typically used when delivering CBT-I in a face-to-face format, following the same general structure: 1) Core objectives (what will be learned and why this information is important), 2) review of previous week's homework and sleep diary data, 3) new intervention material, 4) assignment of homework (treatment strategies for the coming week), and 5) a summary of the Core's main points. Intervention content is enhanced through a variety of interactive features, including personalized goal-setting, graphical feedback based on inputted symptoms, animations / illustrations to enhance comprehension, quizzes to test user knowledge, patient vignettes, and video-based expert explanation. Automated emails are also sent to encourage program adherence. There is no content that is specifically about cancer or caregiving.

Caregivers participating in this study will complete a baseline assessment (questionnaires and 2 weeks of daily sleep diaries), and then will receive complementary and voluntary access to SHUTi. Participants who choose to complete 1 or more SHUTi Cores will complete a follow-up assessment of questionnaires and 2 weeks of sleep diaries; participants who choose not to complete any SHUTi cores will be asked to provide brief feedback regarding their reasons/barriers.

ELIGIBILITY:
Inclusion Criteria:

* self-report providing unpaid care (e.g., practical, medical, and/or emotional support) to an adult family member or "family-like" close individual who is either currently undergoing any anti-cancer treatment (e.g., surgery, chemotherapy, radiation, for either curative or palliative intent) or has completed anti-cancer treatment within the past 2 years.
* Insomnia severity index score of 10 or higher
* age 18 and over
* regular access (at least 2/week) and willingness to use a computer and the Internet and check email
* ability to read and speak English
* resident of the US

Exclusion Criteria:

* irregular sleep schedules that prevent the ability to follow intervention recommendations (i.e., with usual bedtimes outside of 8:00pm to 2:00am or arising time outside of 4:00am to 10:00am)
* current psychological treatment for insomnia
* screen positive for a history of psychotic or bipolar disorder; and current severe depression, high risk of suicide, substance use (alcohol, drug) disorder within the past year
* symptoms suggestive of untreated sleep disorders other than insomnia (e.g., obstructive sleep apnea, restless legs syndrome, periodic limb movement disorder)
* presence of uncontrolled medical condition that is deemed to interfere with the study procedures, or put the study participant at undue risk
* Unstable medication regimen (change to schedule or dosage within past 3 months) for a prescription medication regimen thought to impact sleep.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
SHUTi Usage | 9 weeks
  Number of SHUTi Cores completed by participants

SECONDARY OUTCOMES:
Insomnia severity | Baseline, 9 weeks
  Insomnia severity index; 7 items; summed scores range from 0 to 28 (higher scores indicate more severe insomnia symptoms)
Sleep onset latency (SOL) | Baseline, 9 weeks
  Data collected from sleep diary: Time fell asleep - Time attempting to fall asleep
Wake after sleep onset (WASO) | Baseline, 9 weeks
  Data collected from sleep diary: Total time awake between time feel asleep and final morning waking
Perceived sleep quality | Baseline, 9 weeks
  Data collected from sleep diary: Nightly rating of perceived sleep quality from very poor to very good
Sleep-related cognitions | Baseline, 9 weeks
  Dysfunctional Beliefs and Attitudes about Sleep; 16 items; averaged scores range from 0 to 10 (higher scores indicate more dysfunctional attitudes and beliefs about sleep)
Sleep self-efficacy | Baseline, 9 weeks
  Sleep Self-Efficacy Scale; 13-items; averaged scores range from 0 to 10 (higher scores indicate greater self-efficacy)
Internal and chance sleep locus of control | Baseline, 9 weeks
  Sleep Locus of Control Scale; 4-item subscales for internal and chance locus of control, respectively; averaged scores per scale range from 1 to 6 (higher scores indicate higher belief in the locus of control measured)
Caregiving burden | Baseline, 9 weeks
  Pearlin Stress Scale - Overload subscale; 4 items; averaged scores range from 1 to 4 (higher scores indicate greater perceived burden)
Caregiving competence | Baseline, 9 weeks
  Pearlin Stress Scale - Caregiving Competence subscale; 4 items; averaged scores range from 1 to 4 (higher scores indicate greater perceived competence)
Physical Function | Baseline, 9 weeks
  PROMIS SF v2.0 - Physical Function 8b; 8 items; scored on a normalized T-score distribution (higher scores indicate higher physical function)
Anxiety | Baseline, 9 weeks
  PROMIS SF v2.0 - Anxiety 8a; 8 items; scored on a normalized T-score distribution (higher scores indicate higher anxiety)
Depression | Baseline, 9 weeks
  PROMIS SF v2.0 - Depression 8a; 8 items; scored on a normalized T-score distribution (higher scores indicate higher depression)
Fatigue | Baseline, 9 weeks
  PROMIS SF v2.0 - Fatigue 8a; 8 items; scored on a normalized T-score distribution (higher scores indicate higher fatigue)
Sleep Disturbance | Baseline, 9 weeks
  PROMIS SF v2.0 - Sleep Disturbance 8a; 8 items; scored on a normalized T-score distribution (higher scores indicate higher sleep disturbance)
Social functioning | Baseline, 9 weeks
  PROMIS SF v2.0 - Ability to Participant in Social Roles and Activities 8a; 8 items; scored on a normalized T-score distribution (higher scores indicate higher social function)
Pain Interference | Baseline, 9 weeks
  PROMIS SF v2.0 - Pain Interference 8a; 8 items; scored on a normalized T-score distribution (higher scores indicate higher pain interference)
Pain Intensity | Baseline, 9 weeks
  PROMIS SF v2.0 - Pain Intensity item; 1 item (higher score indicate higher pain intensity)
Experiences with Internet intervention | 9 weeks
  Internet Intervention Utility Questionnaire (UQ) for SHUTi; 18 items; items examined individually
Perceptions of Internet intervention | 9 weeks
  Internet Intervention Impact and Effectiveness Questionnaire (IEQ) for SHUTi; 29 items; items examined individually
Adherence to Internet intervention | 9 weeks
  Internet Intervention Adherence Questionnaire (AQ) for SHUTi; 20 items; items examined individually
SHUTi Feasibility as assessed by open-ended feedback | 9 weeks
  Open-ended survey items regarding barriers to using SHUTi
SHUTi Acceptability as assessed by open-ended feedback | 9 weeks
  Open-ended survey items regarding appropriateness of SHUTi to address caregivers' sleep needs

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Shaffer, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Ritterband LM, Thorndike FP, Ingersoll KS, Lord HR, Gonder-Frederick L, Frederick C, Quigg MS, Cohn WF, Morin CM. Effect of a Web-Based Cognitive Behavior Therapy for Insomnia Intervention With 1-Year Follow-up: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jan 1;74(1):68-75. doi: 10.1001/jamapsychiatry.2016.3249. PMID 27902836
- [Background] Shaffer KM, Garland SN, Mao JJ, Applebaum AJ. Insomnia among Cancer Caregivers: A Proposal for Tailored Cognitive Behavioral Therapy. J Psychother Integr. 2018 Sep;28(3):275-291. doi: 10.1037/int0000105. PMID 30245560
- See also: Center for Behavioral Health and Technology website — https://med.virginia.edu/bht/